CLINICAL TRIAL: NCT05635981
Title: Effect of an Additional Hydrophobic Adhesive Layer Application on the Clinical Performance of Class V Composite Restorations: an 18-month Randomized Clinical Trial
Brief Title: Effect of an Additional Hydrophobic Adhesive Layer Application on the Class V Composite Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meric Berkman, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/76
Record Dates: First submitted 2022-10-28; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Non Carious Cervical Lesion
Keywords: Non Carious Cervical Lesion; Additional Adhesive Layer Application; FDI Criteria; Class V Restorations; Split-Mouth Clinical Study

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The operator who performed the composite restorations is not blinded. Two evaluators who are responsible for the assessment of the clinical performance of restorations according to FDI criteria and the participants are blinded to the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Clearfil S3 Bond Plus (Active Comparator): After selective etching is applied to the enamel surface, Clearfil S3 Bond Plus is applied according to the manufacturer's instructions, restorations are completed with Clearfil Majesty ES-2.
  Clearfil S3 Bond Plus: one-step self-etch adhesive with HEMA
  Interventions: Other: Clearfil Majesty ES-2 Resin Composit Application to Non-carious Cervical Lesions
- Clearfil S3 Bond Plus with Additional Hydrophobic Adhesive Layer Application (Experimental): After selective etching is applied to the enamel surface, Clearfil S3 Bond Plus is applied according to the manufacturer's instructions. Heliobond is applied as an additional hydrophobic adhesive layer and restorations are completed with Clearfil Majesty ES-2.
  Clearfil S3 Bond Plus: one-step self-etch adhesive with HEMA Heliobond: hydrophobic adhesive with Bis-GMA and TEGDMA
  Interventions: Other: Clearfil Majesty ES-2 Resin Composit Application to Non-carious Cervical Lesions
- G-Premio Bond (Active Comparator): After selective etching is applied to the enamel surface, G-Premio Bond is applied according to the manufacturer's instructions, restorations are completed with Clearfil Majesty ES-2.
  G-Premio Bond: universal adhesive without HEMA
  Interventions: Other: Clearfil Majesty ES-2 Resin Composit Application to Non-carious Cervical Lesions
- G-Premio Bond with Additional Hydrophobic Adhesive Layer Application (Experimental): After selective etching is applied to the enamel surface, G-Premio Bond is applied according to the manufacturer's instructions. Heliobond is applied as an additional hydrophobic adhesive layer and restorations are completed with Clearfil Majesty ES-2.
  G-Premio Bond: universal adhesive without HEMA Heliobond: hydrophobic adhesive with Bis-GMA and TEGDMA
  Interventions: Other: Clearfil Majesty ES-2 Resin Composit Application to Non-carious Cervical Lesions

INTERVENTIONS:
Other: Clearfil Majesty ES-2 Resin Composit Application to Non-carious Cervical Lesions — A restorative treatment method that is applied to non-carious cervical lesions using composite resin restoration after adhesive material application.

SUMMARY:
In restorative dentistry, to enhance bond strength between dentin and simplified adhesive systems, new materials or applications are constantly being developed all the time. In order to create a better hybrid layer quality, modifications are made to the chemical contents and application methods of the adhesives. For inhibition or slow down of collagen or resin matrix degradation at the adhesive interface, procedures like using protease enzyme inhibitors or additional hydrophobic layer applications are tested by in vitro and in vivo studies.

The main goal of this double-blind randomized clinical trial is to evaluate the 18-month clinical performances of two different one-step dentin adhesives that were applied alone or with an additional hydrophobic adhesive layer to non-carious cervical lesions.

The hypotheses are that (1) Additional Hydrophobic Adhesive layer application can provide better clinical performance in class V restorations and, (2) the HEMA content will cause statistically different clinical performances.

DETAILED DESCRIPTION:
In this study, Clearfil S3 Bond Plus (one-step self-etch adhesive), G-Premio Bond (Universal adhesive), Heliobond (additional hydrophobic adhesive), and Clearfil Majesty ES-2 (nano-hybrid composite) materials will be used. After performing selective etching with Scotchbond Universal Etchant, four different adhesive procedures will be applied according to manufacturers' instructions to the non-carious cervical lesions selected by the randomized method. In the first group Clearfil S3 Bond Plus, in the second group Clearfil S3 Bond Plus and additional hydrophobic adhesive layer (Heliobond), in the third group G-Premio Bond, in the fourth group, G-Premio Bond and additional hydrophobic adhesive layer (Heliobond) will be applied to the NCCL lesions. Restorations will be accomplished by using Clearfil Majesty ES-2 composite material. Restorations will be evaluated according to FDI criteria. Esthetic properties will be evaluated with surface luster, marginal staining, color match and translucency, esthetic anatomical form parameters. Functional properties will be evaluated with fracture and retention, and marginal adaptation parameters. Biological properties will be evaluated with post-operative sensitivity, periodontal response, and secondary caries parameters. Scores 1, 2, and 3 represent clinically acceptable restorations, and scores 4 and 5 represent clinically unacceptable restorations.

ELIGIBILITY:
Inclusion Criteria:

* 18 and over 18 years old
* Having acceptable oral hygiene
* Good general health
* Having at least 20 teeth in occlusion
* Presence of at least 4 non-carious cervical lesions in the mouth that require treatment
* Lesions without caries
* Patient's consent to come to control appointments
* Vital and non-mobility of the tooth with the lesion
* During occlusion, the tooth with the lesion is in contact with the antagonist tooth.

Exclusion Criteria:

* Under 18 years old
* Having poor oral hygiene
* Poor general health condition
* Pregnancy or breastfeeding status
* Orthodontic application in the last 3 months
* The tooth with the lesion has pulpitis, mobility or it is non-vital
* Presence of advanced bruxism
* The tooth with the lesion is a prosthetic abutment
* Presence of advanced periodontitis or periodontal surgery in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Fracture and Retention | 18 month
  While scoring the fracture and retention parameters, restoration; If there is no fracture with a score of 1 if there are linear cracks with a score of 2 if there are large cracks and fractures that do not affect the marginal integrity and contact with a score of 3 if there are small fractures affecting the marginal integrity or contact or if there are fractures less than half the size of the restoration a score of 4 is a large part of the restoration or In case of losing all, it is evaluated with a score of 5.
Surface Luster | 18 month
  Restoration; A score of 1 if the surface's glossiness is at the same level as enamel, a score of 2 if there are opacity and pores that cannot be noticed from the speaking distance, an acceptable opacity when covered with saliva, or a score of 3 if more than 1/3 of the surface has pores, and a score of 4 if there is a roughness that cannot be masked with saliva and cannot be removed by polishing. If there is a roughness that causes plaque retention, it is evaluated with a score of 5.
Marginal Staining | 18 month
  It is scored as 1 if there is no discoloration on the marginal edges, 2 if there is discoloration that can be easily removed by polishing, 3 if there is moderate discoloration that cannot be accepted aesthetically, 4 if there is noticeable large discoloration that requires repair, and 5 if there is deep marginal discoloration that cannot be repaired.
Marginal Adaptation | 18 month
  If there is no gap at the marginal margins and the tooth tissue is compatible 1, if there is a small gap, line, fracture or step that can be removed by polishing, 2 if there are indentations, if there is a small gap that cannot be removed by polishing, if there is more than one marginal fracture or large indentations 3, if the dentin is exposed repair It is scored 4 if there are large openings, fractures, or indentations that require it, and 5 if there are large openings and irregularities where part of the restoration is lost.
Color Match and Translucency | 18 month
  While scoring the color match and translucency, the restoration and the tissue color are compatible with each other and there is no difference in translucency 1, if there are minor changes in color or translucency 2, if there is a clear but acceptable color difference (more opaque-translucent-light-dark) 3, at a level that can be corrected with repair and 4 if there is a significant color difference, and 5 if there is an unacceptable color difference.
Esthetic Anatomical Form | 18 month
  While scoring the aesthetic anatomical form, the form of the restoration is scored 1 if it is ideal, 2 if it is not ideal but will be ideal with a small intervention, 3 if it is not ideal but aesthetically acceptable, 4 if it is not aesthetically acceptable and repair is required, and 5 if it is unacceptable and needs to be changed.
Periodontal Response | 18 month
  During periodontal response scoring, if there is no plaque accumulation, pocket formation or inflammation in the restored tooth, 1, if there is a small amount of plaque accumulation and no inflammation and pocket formation, 2, if the papillary bleeding index increases by 1 point compared to the baseline, 3 if the papillary bleeding index increases by more than 1 point and periodontal bleeding index increases by more than 1 point It is scored 4 if there is an increase in the pocket more than 1 mm, and 5 if there is acute gingivitis or acute periodontitis.
Post Operative Sensitivity | 18 month
  Restoration; It is evaluated with a score of 1 if there is no sensitivity complaint, with a score of 2 if there is a small amount of sensitivity for a short time, and a score of 3 if the patient has no complaints and moderate sensitivity, with a score of 3 if there is hypersensitivity that does not require restoration replacement but requires repair, and a score of 4 if endodontic treatment is required.
Secondary Caries | 18 month
  Restoration; It is evaluated with a score of 1 if there is no caries formation, with a score of 2 if there is small and localized demineralization, and a score of 3 if there is demineralization in a large area that requires only precautions, and a score of 4 if there is cavitation that requires repair, and a score of 5 if there is a deep caries that cannot be repaired.

CONTACTS AND LOCATIONS:
Overall Officials: Meriç Berkman, pHD, Principal Investigator — Istanbul University; Safa Tuncer, Professor, Study Chair — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code